CLINICAL TRIAL: NCT01399957
Title: Responsiveness to Dalfampridine Treatment Among Multiple Sclerosis Patients Followed at the Mandell MS Center: Characterizing Clinical Predictors of Response and Identifying Additional Outcomes
Brief Title: Responsiveness to Dalfampridine-ER Treatment Among Multiple Sclerosis Patients
Status: Completed | Type: Observational
Sponsor: Mount Sinai Rehabilitation Hospital (Other)
Collaborators: Brown University (Other); Acorda Therapeutics (Industry)
Responsible Party: Principal Investigator, Jennifer Ruiz, DPT, Research Manager, Mount Sinai Rehabilitation Hospital
Other Study IDs: AL0003
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Dalfampridine-ER; Walking speed
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 15 mL of blood will be collected into an EDTA tube from participants at assessment appointments. Both serum and cells will be frozen and stored in a -80 degree freezer.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pwMS prescribed dalfampridine-ER: Anyone prescribed D-ER per usual clinical care was recruited into this observational study. All those willing to participate were consented and observed pre-drug and for a 14week period with two follow-up visits scheduled at 12 and 18months.

SUMMARY:
Ampyra (dalfampridine-ER) was approved by the FDA (2010) for improving walking speed in persons with multiple sclerosis. This project seeks to determine if there are other benefits to taking dalfampridine besides an increase in walking speed. This is strictly an observational study and research staff will not be involved in any decisions to stop or start taking the medication.

DETAILED DESCRIPTION:
Subjects will be evaluated before starting medication, throughout a 14week period after starting D-ER as well as at 12 and 18months following the start date of medication regardless of if they stayed on medication or not.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of MS by McDonald criteria
* Prescribed ampyra (dalfampridine) as part of usual care, but have not yet started taking the medication before baseline visit
* Receive MS care at the Mandell MS center
* Cognitively able to understand directions and complete protocol (score of 22 or greater on the MMSE)
* 18 years of age or older

Exclusion Criteria:

* Already began to take drug prior to baseline research visit
* Not planning to continue care at Mandell Center for at least 14 weeks after initiation of therapy
* Unwilling or unable to complete assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with MS who have been prescribed ampyra at the Mandell Center for Multiple Sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2010-08; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in 25ft walk time | Baseline (pre drug) and followup at 3.5 weeks, 7 weeks, 10.5 weeks and 14weeks
Change in 6 minute walk distance | Baseline (pre drug) and followup at 3.5 weeks, 7 weeks, 10.5 weeks and 14weeks
  Measure of endurance

SECONDARY OUTCOMES:
Change of Upper extremity dexterity with 9hole peg test | Baseline (pre drug) and followup at 3.5 weeks, 7 weeks, 10.5 weeks and 14weeks

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lo, M.D, Ph.D., Principal Investigator — Mandell Center for Multiple Sclerosis at Mount Sinai Rehabilitation Hospital; Elizabeth Triche, Ph.D, Principal Investigator — Brown University
Locations (1):
- Mandell Center for Multiple Sclerosis at the Mount Sinai Rehabilitation Hospital, Hartford, Connecticut, United States